CLINICAL TRIAL: NCT00420875
Title: "Clinical Evaluation of Placement of Radiofrequency-based Plasma Microdebridement in the Treatment Algorithm for Foot and Ankle Tendinosis and Plantar Fasciosis"
Brief Title: Clinical Evaluation of Placement of Radiofrequency-based Plasma Microdebridement in the Treatment Algorithm for Foot and Ankle Tendinosis and Plantar Fasciosis
Acronym: TOPAZ Registry
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not meet enrollment goals
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Dr. Tara Waterman, Director of Medical Affairs, ArthroCare Corporation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM-706WW
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Plantar Fasciosis, Achilles Tendinosis
Keywords: plantar fasciitis; plantar fasciosis; Achilles tendinosis; Achilles tendinitis; heel pain; fasciosis; fasciitis; tendinosis; tendinitis; conservative treatment
MeSH Terms: conditions — Fasciitis, Plantar; Fasciitis; Tendinopathy

INTERVENTIONS:
Device: TOPAZ MicroDebrider — The TOPAZ MicroDebrider will be used for patients that fail conservative care. Under sterile conditions in the operating room, patients will be given intravenous sedation (drugs that make you sleepy and unaware of your surroundings) in a hand vein and local anesthetic (drugs to numb the area where the surgical procedure will be done). Depending on the technique used the study doctor may or may not make an incision (cut) about 1 inch long on the side of your foot to expose your tendon. If the study doctor chooses to use the percutaneous method, an incision will not be made. The study doctor will put the tip of the TOPAZ MicroDebrider device (which is about 1/16th of an inch long) into the tendon. A current of energy will be applied on and around the tendon. Steri strips will be placed on the skin to close the area treated.

SUMMARY:
To determine the magnitude of improvement for pain and function symptoms over a two year period after enrollment into the registry study in patients presenting with chronic heel pain and receiving standard of care treatment. Standard of care will include traditional conservative care measures, ESWT, radiofrequency-based plasma microdebridement, scalpel debridement and/or surgical release.

DETAILED DESCRIPTION:
Several million Americans receive treatment for heel pain each year, with more than two million patients treated each year for plantar fasciitis and fasciosis alone.(2) Conservative treatment options for recalcitrant heel pain include rest, stretching, strengthening and massage, progressing to non-steroidal anti-inflammatory drugs (NSAIDs), cox-2 inhibitors, steroid injections or iontophoresis with continued recalcitrance.(3;4) Orthotics, heel cups, night splints and plantar strapping are other conservative options frequently recommended by treating physicians.(4) Patient outcomes and response to conservative measures is usually positive, with non-responsive cases, approximately 2% - 10% of all presenting cases, receiving surgical care. Extracorporeal shockwave treatment (ESWT) has recently been advocated for the recalcitrant cases and has shown to be effective in 60-80 percent of the cases.(5-7) In general, non-surgical treatment of plantar fasciosis and tendinosis is believed to be unsuccessful, so that surgical treatment is required in about 25% of patients; however, results of traditional surgical treatments have been reported to deteriorate with time.(8)

Clinical experience following RF-based plasma microtenotomy has demonstrated excellent success in treating chronic, refractive tendinosis of the lateral epicondyle in the elbow.(9) The investigators reported that this technique was technically simple to perform and was much less invasive than conventional surgery. Patients had a rapid and uncomplicated recovery and reported minimal to no pain 7-10 days following the procedure; their pain relief persisted or improved through 24 months. Magnetic resonance imaging correlated well with clinical results. The RF-based plasma microtenotomy procedure is also being used successfully in tendons in the shoulder, knee, foot and ankle and in the plantar fascia. A randomized controlled study was conducted with the aim of determining whether bRF-based microtenotomy was effective for treating chronic supraspinatus tendinosis (10). Longitudinal postoperative recovery through one year for patients treated using RF-based plasma microtenotomy was compared to patients undergoing subacromial decompression. Both patient groups demonstrated significant improvement after each respective procedure and longitudinal recovery profiles were statistically similar. Early experience using this procedure for foot and ankle tendons, including the Achilles tendon, posterior tibial tendon, peroneal tendon, and plantar fascia revealed over 90% good to excellent results, reflecting the results shown by patients treated for tendinosis in the elbow (11)

Further investigation of optimal placement of this surgical approach into the standard of care treatment paradigm for treating plantar fasciosis and Achilles tendinosis would be beneficial. It is not known whether this RF-based plasma microsurgery might be more optimally placed earlier on within the standard of care treatment algorithm.

The purpose of this study is to determine the magnitude of improvement for pain and functional symptoms over a two year period after enrollment into the registry study in patients presenting with chronic heel pain and undergoing standard of care treatment. Standard of care will include traditional conservative care measures, ESWT, radiofrequency-based plasma microdebridement, scalpel debridement and/or surgical release.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject's history and physical examination pinpoints anatomic origin of heel pain as associated with plantar fasciosis (tenderness with palpation and local pressure over the medial calcaneal tuberosity on passive dorsiflexion) or Achilles tendinosis (tenderness upon palpation and local pressure at the insertion site)
* Subject (or guardian) must sign IRB approved informed consent form
* Subject is willing and able to complete required follow-up

Exclusion Criteria:

* Previous fascia surgery on pathology to be treated by this study
* Multiple anatomic origins of heel pain in foot to be treated by study
* History or documentation showing Type I and Type II Diabetes Mellitus
* Physical findings and documentation of coagulopathy, infection, tumor or other systemic disease(s)
* History or documentation showing peripheral vascular disease or autoimmune disease
* History or documentation of fibromyalgia
* Subject is currently participating in another drug/device study related to the injured plantar fascia or Achilles tendon
* Pregnant or pregnant suspected subjects prior to treatment
* Subject is incapable of understanding or responding to the study questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Ankle Hind Foot Scale (AHS) | 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months

SECONDARY OUTCOMES:
Visual Analog Scale (VAS), SF-36 Quality of Life, Patient Satisfaction | 6 weeks, 3 months, 6 months, 12 months, 18 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Babak Baravarian, DPM, Principal Investigator — Foot and Ankle Institute of Santa Monica
Locations (3):
- United States (3):
  - Foot Care Physicians, Mesa, Arizona
  - Foot and Ankle Institute of Santa Monica, Santa Monica, California
  - Foot and Ankle Clinic of Oakwood, Oakwood, Georgia

REFERENCES:
- [Background] Aldridge T. Diagnosing heel pain in adults. Am Fam Physician. 2004 Jul 15;70(2):332-8. PMID 15291091
- [Background] Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID 12756315
- [Background] Yu JS. Pathologic and post-operative conditions of the plantar fascia: review of MR imaging appearances. Skeletal Radiol. 2000 Sep;29(9):491-501. doi: 10.1007/s002560000230. PMID 11000294
- [Background] LeMelle DP, Kisilewicz P, Janis LR. Chronic plantar fascial inflammation and fibrosis. Clin Podiatr Med Surg. 1990 Apr;7(2):385-9. PMID 2346891
- [Background] Schepsis AA, Leach RE, Gorzyca J. Plantar fasciitis. Etiology, treatment, surgical results, and review of the literature. Clin Orthop Relat Res. 1991 May;(266):185-96. PMID 2019049
- [Background] Strash WW, Perez RR. Extracorporeal shockwave therapy for chronic proximal plantar fasciitis. Clin Podiatr Med Surg. 2002 Oct;19(4):467-76. doi: 10.1016/s0891-8422(02)00016-2. PMID 12471854
- [Background] Lewis G, Gatti A, Barry LD, Greenberg PM, Levenson M. The plantar approach to heel surgery: a retrospective study. J Foot Surg. 1991 Nov-Dec;30(6):542-6. PMID 1770205
- [Background] Regan W, Wold LE, Coonrad R, Morrey BF. Microscopic histopathology of chronic refractory lateral epicondylitis. Am J Sports Med. 1992 Nov-Dec;20(6):746-9. doi: 10.1177/036354659202000618. PMID 1280910
- [Background] Goldberg EJ, Abraham E, Siegel I. The surgical treatment of chronic lateral humeral epicondylitis by common extensor release. Clin Orthop Relat Res. 1988 Aug;(233):208-12. PMID 3402125
- [Background] Galliani I, Burattini S, Mariani AR, Riccio M, Cassiani G, Falcieri E. Morpho-functional changes in human tendon tissue. Eur J Histochem. 2002;46(1):3-12. doi: 10.4081/1649. PMID 12044045
- [Background] Nirschl RP, Ashman ES. Elbow tendinopathy: tennis elbow. Clin Sports Med. 2003 Oct;22(4):813-36. doi: 10.1016/s0278-5919(03)00051-6. PMID 14560549
- [Background] Stone PA, McClure LP. Retrospective review of endoscopic plantar fasciotomy. 1994 through 1997. J Am Podiatr Med Assoc. 1999 Feb;89(2):89-93. doi: 10.7547/87507315-89-2-89. PMID 10063779
- [Background] Gould JS. Chronic plantar fasciitis. Am J Orthop (Belle Mead NJ). 2003 Jan;32(1):11-3. No abstract available. PMID 12580344
- [Background] Hammer DS, Adam F, Kreutz A, Rupp S, Kohn D, Seil R. Ultrasonographic evaluation at 6-month follow-up of plantar fasciitis after extracorporeal shock wave therapy. Arch Orthop Trauma Surg. 2005 Feb;125(1):6-9. doi: 10.1007/s00402-003-0591-z. Epub 2003 Oct 3. PMID 14530990
- [Background] Hyer CF, Vancourt R, Block A. Evaluation of ultrasound-guided extracorporeal shock wave therapy (ESWT) in the treatment of chronic plantar fasciitis. J Foot Ankle Surg. 2005 Mar-Apr;44(2):137-43. doi: 10.1053/j.jfas.2005.01.005. PMID 15768363
- [Background] Theodore GH, Buch M, Amendola A, Bachmann C, Fleming LL, Zingas C. Extracorporeal shock wave therapy for the treatment of plantar fasciitis. Foot Ankle Int. 2004 May;25(5):290-7. doi: 10.1177/107110070402500503. PMID 15134608
- [Background] Alfredson H, Lorentzon R. Chronic Achilles tendinosis: recommendations for treatment and prevention. Sports Med. 2000 Feb;29(2):135-46. doi: 10.2165/00007256-200029020-00005. PMID 10701715
- [Background] Hardy RI, James FW, Millard RW, Kaplan S. Regional myocardial blood flow and cardiac mechanics in dog hearts with CO2 laser-induced intramyocardial revascularization. Basic Res Cardiol. 1990 Mar-Apr;85(2):179-97. doi: 10.1007/BF01906971. PMID 2350332
- [Background] Hughes GC, Biswas SS, Yin B, Baklanov DV, Annex BH, Coleman RE, DeGrado TR, Landolfo CK, Landolfo KP, Lowe JE. A comparison of mechanical and laser transmyocardial revascularization for induction of angiogenesis and arteriogenesis in chronically ischemic myocardium. J Am Coll Cardiol. 2002 Apr 3;39(7):1220-8. doi: 10.1016/s0735-1097(02)01734-5. PMID 11923050
- [Background] Horvath KA, Belkind N, Wu I, Greene R, Doukas J, Lomasney JW, McPherson DD, Fullerton DA. Functional comparison of transmyocardial revascularization by mechanical and laser means. Ann Thorac Surg. 2001 Dec;72(6):1997-2002. doi: 10.1016/s0003-4975(01)03243-x. PMID 11789783
- [Background] Dietz U, Horstick G, Manke T, Otto M, Eick O, Kirkpatrick CJ, Meyer J, Darius H. Myocardial angiogenesis resulting in functional communications with the left cavity induced by intramyocardial high-frequency ablation: histomorphology of immediate and long-term effects in pigs. Cardiology. 2003;99(1):32-8. doi: 10.1159/000068450. PMID 12589120
- [Background] Fisher PE, Khomoto T, DeRosa CM, Spotnitz HM, Smith CR, Burkhoff D. Histologic analysis of transmyocardial channels: comparison of CO2 and holmium:YAG lasers. Ann Thorac Surg. 1997 Aug;64(2):466-72. doi: 10.1016/S0003-4975(97)00519-5. PMID 9262595
- [Background] Kohmoto T, DeRosa CM, Yamamoto N, Fisher PE, Failey P, Smith CR, Burkhoff D. Evidence of vascular growth associated with laser treatment of normal canine myocardium. Ann Thorac Surg. 1998 May;65(5):1360-7. doi: 10.1016/s0003-4975(98)00236-7. PMID 9594867
- [Background] Kwon HM, Hong BK, Jang GJ, Kim DS, Choi EY, Kim IJ, McKenna CJ, Ritman EL, Schwartz RS. Percutaneous transmyocardial revascularization induces angiogenesis: a histologic and 3-dimensional micro computed tomography study. J Korean Med Sci. 1999 Oct;14(5):502-10. doi: 10.3346/jkms.1999.14.5.502. PMID 10576145
- [Background] Yamamoto N, Gu A, DeRosa CM, Shimizu J, Zwas DR, Smith CR, Burkhoff D. Radio frequency transmyocardial revascularization enhances angiogenesis and causes myocardial denervation in canine model. Lasers Surg Med. 2000;27(1):18-28. doi: 10.1002/1096-9101(2000)27:13.0.co;2-f. PMID 10918289
- [Background] O'Neill CW, Liu JJ, Leibenberg E, Hu SS, Deviren V, Tay BK, Chin CT, Lotz JC. Percutaneous plasma decompression alters cytokine expression in injured porcine intervertebral discs. Spine J. 2004 Jan-Feb;4(1):88-98. doi: 10.1016/s1529-9430(03)00423-6. PMID 14749197
- [Background] Tasto JP, Cummings J, Medlock V, Hardesty R, Amiel D. Microtenotomy using a radiofrequency probe to treat lateral epicondylitis. Arthroscopy. 2005 Jul;21(7):851-60. doi: 10.1016/j.arthro.2005.03.019. PMID 16012499
- [Background] Leitze Z, Sella EJ, Aversa JM. Endoscopic decompression of the retrocalcaneal space. J Bone Joint Surg Am. 2003 Aug;85(8):1488-96. doi: 10.2106/00004623-200308000-00009. PMID 12925628
- [Background] Buttermann GR. Treatment of lumbar disc herniation: epidural steroid injection compared with discectomy. A prospective, randomized study. J Bone Joint Surg Am. 2004 Apr;86(4):670-9. PMID 15069129
- [Background] Sharps LS, Isaac Z. Percutaneous disc decompression using nucleoplasty. Pain Physician. 2002 Apr;5(2):121-6. PMID 16902662
- [Background] Singh V, Piryani C, Liao K, Nieschulz S. Percutaneous disc decompression using coblation (nucleoplasty) in the treatment of chronic discogenic pain. Pain Physician. 2002 Jul;5(3):250-9. PMID 16902650
- See also: Click here for information about TOPAZ (the device to be used in the study) — http://topazinfo.com